CLINICAL TRIAL: NCT03865823
Title: Evaluation of the Recovery Rate and Postoperative Incontinence of Surgical Fistulas in a Cohort of a Reference Centre
Acronym: PROFIL
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Other Study IDs: D_ELK_2018_2
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anal Fistula
Keywords: anal fistula; anal infection
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- anal Fistula: patient with anal fistula with indication to surgical treatment
  Interventions: Procedure: pus sample

INTERVENTIONS:
Procedure: pus sample — A pus sample from the fistula will be taken by the doctor during this first consultation or, failing that, in the operating room before disinfection.

SUMMARY:
Fistula is a pathology that can be complex and lead to treatment difficulties for the proctologist.

The proctologist's objective is to treat the infection (anal fistula and abscess) with the minimum impact on anal continence. Drainage of the fistula pathway(s) and removal of infected tissue during initial surgery are essential. The treatment of upper trans-sphincterial fistulas, i. e. those that span more than half the height of the anal sphincter, poses risks to anal continence. It sometimes requires several times of surgical treatment.

The study aim to investigate the fate of all patients treated for anal fistula in an expert team, in terms of impact on healing and anal continence and according to the type of anal fistula, the co-morbidity, the surgical techniques used and the bacterial flora responsible.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18, patient with an anus fistula with indication for surgical treatment

Exclusion Criteria:

* Cutaneous Suppuration, without fistula (e.g., Verneuil disease, boil)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an anus fistula with indication for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Healing rate at 2 years after initial surgical management of anal fistula. | 2 years
  Healing is defined by the absence of anal pain, pus discharge and anal swelling reported by the patient.

SECONDARY OUTCOMES:
Anal incontinence rate in participants operated for anal fistula, 2 years after initial care. | Year 2
  Rate of anal incontinence and degree of continence impairment assessed by the change in the Vaizey score preoperatively and postoperatively at 2 years after initial treatment.
  Anal incontinence is defined by a Vaizey score > 4 reported by the participant during a phone interview. The Vaizey score ranges from 0 to 24/24, with the higher the score, the greater the loss of continence. Perfect continence therefore corresponds to 0/24. Normal" continence can be defined as continence ranging from 0 to 4/24.
Healing rate in participants operated for anal fistula, at 6, 12 and 24 months after initial care. | Month 6, 12, 24
  Healing is defined by the absence of anal pain, pus discharge and anal swelling reported by the patient at 6, 12 and 24 months.
Assessment of time to consolidated recovery. | Month 24
  Time (in days) between the start of treatment (date of the first operation) and the 'end of follow-up' consultation, at which the surgeon considers the participant to be cured (consolidated cure).
  Consolidated healing is defined by the surgeon:
  * On examination, by the absence of anal pain, pus discharge and anal swelling reported by the participant.
  * On clinical examination, by the complete closure of the scar with re-epithelialisation and the absence of pus discharge.
Description of the number of surgeries required to obtain a cure. | 2 years
  Description of the number and type of anal fistula surgeries performed during the participant's follow-up, at 6, 12 and 24 months.
Bacteriological profile at the level of the fistula at the time of diagnosis and research into a possible role in the cure rate, the surgical technique used and the rate of post-operative incontinence. | 2 weeks
  Description of the bacteriological profile found in the fistula when the pus was sampled at the time of the first consultation or, if this could not be done, when a sample was taken in the operating theatre before starting the surgical procedure.
Quality of life of participants at 2 years. | 2 years
  Changes in quality of life after surgical treatment will be assessed at 6, 12 and 24 months using the FIQL (Fecal Incontinence Quality of Life) score.
  The FIQL questionnaire comprises 29 items grouped into four dimensions: lifestyle, behaviour, depression and self-image, and embarrassment in relation to others. Each item was given a score from 1 to 4 (1 being the worst).
Quantitative assessment of sphincter function using anorectal manometry | 2 years
  Evolution of anal sphincter pressure measurements in people at risk or developing incontinence during follow-up, measured by anorectal manometry: resting pressure below 60mmHg, maximum and mean voluntary contraction in mmHg, length of canal in mm, maximum tolerated volume and perception threshold in ml.
Evolution of anatomical lesions of the anal sphincter on endoanal ultrasound | 2 years
  Evolution of lesions on EndoAnal Ultrasound measured before the first surgery and at 24 months in patients at risk or developing incontinence during follow-up (defined by a worsening of the Vaizey score greater than 4/24) Description of lesions: Presence of a collection with its size (defined as a heterogeneous hypoechoic area with hyperechoic spot, measured in mm, length of the anal fistula in mm, description of the type of fistula (trans-sphincter, inter-sphincter or horseshoe, anterior, posterior, right, left). Measurement of defects in terms of angle, height and volume, specifying internal sphincter, external sphincter and puborectal strap (Stark classification).

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, France

IPD SHARING:
Plan to Share IPD: No